CLINICAL TRIAL: NCT03740711
Title: Early Left Atrial Venting Versus Conventional Treatment For Left Ventricular Decompression During Venoarterial Extracorporeal Membrane Oxygenation Support (EVOLVE-ECMO Trial)
Brief Title: Early LA Venting During Venoaterial ECMO Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Seok Kim, Clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_2018_0646
Record Dates: First submitted 2018-10-19; First posted 2018-11-14 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation Support; Refractory Pulmonary Edema
Keywords: Cardiogenic shock; Extracorporeal Membrane Oxygenation Support; Left atrial venting
MeSH Terms: conditions — Shock, Cardiogenic; Pulmonary Edema

STUDY DESIGN:
Intervention Model Description: Randomized controlled test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early LA venting (Experimental): When detect B-line on serial lung ultrasound, we will perform early LA venting for improving LV distention in patients with refractory cardiogenic shock who received VA-ECMO support.
  Interventions: Procedure: Left atrial venting
- Conventional LA venting (Active Comparator): When detect refractory pulmonary congestion on chest radiograph or inadequate AV opening on serial echocardiography, we will perform LA venting for improving LV distention in patients with refractory cardiogenic shock who received VA-ECMO support.
  Interventions: Procedure: Left atrial venting

INTERVENTIONS:
Procedure: Left atrial venting — The contralateral femoral vein is assessed with an 7-French(Fr) sheath() and femoral artery is assessed with 5-Fr sheath( ) for fluoroscopic guidance using 5-Fr pig-tail catheter. In some cases trans-esophageal echo is used. The inter-atrial septum in punctured with a standard BRK™tran-septal needle(St. Jude Medical Inc., St. Paul, MN) under direct visualization via an 8-Fr Mullin sheath(St. Jude Medical Inc.). A SAFARI™(Boston Scientific, Galway, Ireland) guidewire is advanced into the LA. An 8-Fr Mullin-sheath is removed and atrial septostomy is performed using 21-Fr dilator. A 17-Fr or 21-Fr Biomedicus Percutaneous Femoral cannula(Medtronic Inc., Minneapolis, MN) is then placed in the LA and was attached to the ECMO circuit using a Y connector.

SUMMARY:
The EVOLVE-ECMO(Early Left Atrial Venting Versus Conventional Treatment For Left VEntricular Decompression During Venoarterial ExtraCorporeal Membrane Oxygenation Support) study is a randomized controlled trial to evaluate the prognostic effect of early LA venting(when detect B-line on serial lung ultrasound) on weaning VA-ECMO support in refractory CS who receive VA-ECMO support. The aim of EVOLVE-ECMO trial is to test the hypothesis that early LA venting would result in a significant reduction in failure of weaning ECMO support in refractory CS.

ELIGIBILITY:
Inclusion Criteria:

* Subject was > 18 years of age.
* Subjects who underwent successful VA-ECMO support
* Subjects with refractory cardiogenic shock who had pulmonary edema confirmed by chest X ray or lung sonogram.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* subject was <80 years of age
* Pregnant and/or lactate women
* Subjects who underwent VA-ECMO after recent open heart surgery
* Subjects who underwent VA-ECMO after non-cardiogenic arrest(trauma, hypothermia, submersion, drug overdose, asphyxia, intracranial hemorrhage etc)
* Severe bleeding tendency
* Terminal malignancy
* Known severe irreversible brain damage
* Subject was unable to provide written informed consent or participate.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
weaning rate of VA-ECMO | during index admission
  Weaning of VA-ECMO support

SECONDARY OUTCOMES:
In hospital mortality | during index admission
Adverse outcome due to LA venting | during index admission
Free days for mechanical ventilation | during index admission
Success rate to heart transplantation | during index admission
rate of improving for pulmonary edema | during index admission

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided